CLINICAL TRIAL: NCT06967025
Title: Ischemic Postconditioning in Acute Stroke Patients Receiving Endovascular Thrombectomy: Mechanistic Exploration Through a Randomized Controlled Pilot Trial
Brief Title: Ischemic Postconditioning in Acute Stroke Patients Receiving Endovascular Thrombectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Ming Wei, Chief Physician, Tianjin Huanhu Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tjhh20249
Record Dates: First submitted 2025-04-16; First posted 2025-05-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2024-09

CONDITIONS: Stroke Acute; Cytoprotection; Ischemic Conditioning
MeSH Terms: conditions — Stroke | interventions — Ischemic Postconditioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular thrombectomy (Active Comparator)
  Interventions: Procedure: Endovascular Thrombectomy
- Ischemic Postconditioning plus Endovascular thrombectomy (Experimental)
  Interventions: Procedure: Ischemic Postconditioning

INTERVENTIONS:
Procedure: Ischemic Postconditioning — Ischemic Postconditioning will consist of 4 cycles of 2-minute cycles of balloon inflation (occlusion) followed by 2 minutes of deflation (reperfusion), and will be initiated immediately upon successful recanalization (eTICI 2b-3) using low pressure balloon in situ of the location of thrombus.
  Arms: Ischemic Postconditioning plus Endovascular thrombectomy
Procedure: Endovascular Thrombectomy — Thrombectomy alone.
  Arms: Endovascular thrombectomy

SUMMARY:
This clinical trial will evaluate whether on-site ischemic postconditioning (IPostC) improves outcomes in acute stroke patients receiving endovascular thrombectomy (EVT) and explore its mechanisms. The investigators aim to answer: (1) Is on-site IPostC effective compared to EVT alone? (2) What molecular markers and cellular pathways does on-site IPostC influence? Participants will be randomized to EVT alone or EVT+IPostC (4 cycles of 2-minute balloon occlusion/reperfusion). The investigators will assess infarct size, functional outcomes, biomarkers (e.g., multi-omics, ELISA, and clinical laboratory parameters), and safety (e.g., mortality, procedure-related complications).

DETAILED DESCRIPTION:
This clinical trial is a single-center, prospective, blind endpoint, randomized -controlled trial. Randomization will be in a 1:1 ratio, Intervention Arm (EVT + on-site IPostC) or Control Arm (EVT alone) in up to a total of 60 patients (30 subjects in each arm). On-site IPostC will be initiated immediately upon successful recanalization (eTICI 2b-3) using low pressure balloon in situ of the location of thrombus, consisting of 4 cycles of 2-minute cycles of balloon inflation (occlusion) followed by 2 minutes of deflation (reperfusion).

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥ 18 years of age.
* The patient must have symptoms consistent with AIS (i.e. face drooping, arm weakness, speech difficulty, etc.) , with symptoms severity of baseline NIHSS ≥ 6 and beginning less than 24 hours prior to presentation at hospital.
* Pre-stroke mRS ≤ 2.
* Baseline ASPECTS ≥ 6.
* Unilateral middle cerebral artery occlusion, and/or internal carotid artery occlusion.
* The patient is eligible for EVT.
* Successful recanalization achieved through EVT (eTICI 2b-3).
* The patient is willing to provide written informed consent to participate in this clinical trial.

Exclusion Criteria:

* The interventionalist deems the study device unable to reach the target site.
* Adverse events related to thrombectomy, such as contrast extravasation, vascular rupture/perforation, dissection, or embolization to a new territory, detected on post-thrombectomy angiography.
* Stent placement performed in the M1 segment of the middle cerebral artery or the terminal segment of the internal carotid artery during thrombectomy.
* Angioplasty of more than two cycles of balloon inflation/deflation.
* The patient is experiencing cardiogenic shock, systolic blood pressure [SBP] <100 mmHg, HR>100 bpm and arterial oxygen saturation (pulse oximetry) <92% without additional oxygen.
* The patient has known history of Congestive Heart Failure, hepatic failure, end-stage kidney disease or severe renal failure (clearance < 30ml/min/1.73m²).
* The patient is febrile (temperature > 37.5 °C) or has experienced an infection with fever in the last 5 days.
* The patient has a known hypersensitivity or contraindication to aspirin, heparin, Clopidogrel, tirofiban, or sensitivity to contrast media, which cannot be adequately pre-medicated.
* The patient has a known history of bleeding diathesis, coagulopathy, cryoglobulinemia, sickle cell anemia, or will refuse blood transfusions.
* The patient has a pre-AIS life expectancy of <1 year due to underlying medical conditions or pre-existing co-morbidities.
* The patient is currently enrolled in another investigational drug or device trial.
* The patient is apprehensive about or unwilling to undergo the required MRI imaging at follow-up, has a documented or suspected diagnosis of claustrophobia, or has Gadolinium allergy.
* The patient is a female who is known to be pregnant.
* Other conditions deemed unsuitable for inclusion by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Infarct volume growth | Difference between infarct volume at 48 (-12/+24) hours post-randomization and baseline.

SECONDARY OUTCOMES:
Final infarct volume | At 48 (-12/+24) hours post-randomization.
Immediate postprocedural infarct volume | Within 2 hours post-randomization.
Difference in modified Rankin Scale distribution | At 90 days post-randomization.
  The modified Rankin Scale (mRS) is a 7-point ordinal scale ranging from 0 (no disability) to 6 (death). Higher scores indicate worse outcomes. The distribution of mRS scores (0-6) will be compared between treatment groups.
Difference in modified Rankin Scale of 0-1 | At 90 days post-randomization.
  The modified Rankin Scale (mRS) is a 7-point ordinal scale ranging from 0 (no disability) to 6 (death). Higher scores indicate worse outcomes. The proportion of mRS 0-1 will be compared between treatment groups.
Difference in modified Rankin Scale of 0-2 | At 90 days post-randomization.
  The modified Rankin Scale (mRS) is a 7-point ordinal scale ranging from 0 (no disability) to 6 (death). Higher scores indicate worse outcomes. The proportion of mRS 0-2 will be compared between treatment groups.
Occurrence of early neurological improvement | within 24 hours post-randomization.
  The National Institutes of Health Stroke Scale (NIHSS) is a 42-point ordinal scale ranging from 0 (no stroke symptoms) to 42 (severe stroke). Higher scores indicate worse neurological deficits. Early neurological improvement is defined as a reduction in NIHSS score by ≥8 points.
Longitudinal Change of NIHSS Scores | At 24 hours, 3 days, and 5-7 days post-randomization or at discharge.
  The National Institutes of Health Stroke Scale (NIHSS) is a 42-point ordinal scale ranging from 0 (no stroke symptoms) to 42 (severe stroke). Higher scores indicate worse neurological deficits. NIHSS scores will be serially assessed at specified intervals.

OTHER OUTCOMES:
Blood brain barrier permeability as measured by K-trans value using dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) | At 48 (-12/+24) hours post-randomization.
Multi-omics analysis of protein and metabolite quantitative changes using mass spectrometry-based proteomics and metabolomics | At 48 (-12/+24) hours post-randomization.
Percentage of platelet-neutrophil aggregates (CD41+CD66b+ cells) measured by flow cytometry | Within 24 hours post-randomization.
Percentage of activated platelets (CD41+CD62+ cells) measured by flow cytometry | Within 24 hours post-randomization.
Percentage of activated neutrophils (CD11b+ cells) measured by flow cytometry | Within 24 hours post-randomization.
R time (reaction time) measured by thromboelastogram (TEG) | Within 24 hours post-randomization.
  Quantitative assessment of clot initiation dynamics using TEG. R time measures the latency to initial fibrin formation (reported in seconds). Lower values indicate faster clot initiation, while higher values suggest delayed clotting.
K time (clot kinetics) measured by thromboelastogram (TEG) | Within 24 hours post-randomization.
  Quantitative assessment of clot formation speed using TEG. K time reflects the time from clot initiation to a fixed clot strength (reported in seconds). Lower values indicate faster clot kinetics, while higher values suggest slower clot formation.
Alpha angle measured by thromboelastogram (TEG) | Within 24 hours post-randomization.
  Quantitative assessment of fibrin polymerization rate using TEG. The alpha angle (reported in degrees) represents the slope of clot strengthening. Higher values indicate faster fibrin cross-linking and clot stability.
MA (maximum amplitude) measured by thromboelastogram (TEG) | Within 24 hours post-randomization.
  Quantitative assessment of clot strength using TEG. MA (reported in millimeters) measures the maximum clot firmness. Higher values indicate stronger clot structure, while lower values suggest weaker clot integrity.
EPL (estimated percent lysis) measured by thromboelastogram (TEG) | Within 24 hours post-randomization.
  Quantitative assessment of clot lysis potential using TEG. EPL (reported as a percentage) estimates the percentage of clot lysed after maximum amplitude is reached. Higher values indicate greater fibrinolysis activity.
LY30 (lysis at 30 minutes) measured by thromboelastogram (TEG) | Within 24 hours post-randomization.
  Quantitative assessment of late-stage clot lysis using TEG. LY30 (reported as a percentage) measures the percentage of clot lysed 30 minutes after maximum amplitude. Higher values indicate increased fibrinolysis over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
Plan Description: De-identified individual participant data (IPD) will not be made publicly available due to unresolved ethical considerations regarding data anonymization feasibility and institutional policies. A formal evaluation of data sharing options will be conducted post-study completion.
  Access Criteria: Not applicable. IPD sharing is currently restricted. Future access may be negotiated via institutional data governance committees upon reasonable request.